CLINICAL TRIAL: NCT02549781
Title: Influence of Sensorimotor Environment on Gambling Behavior in Pathological Gambling.
Brief Title: Environmental Influence on Gambling Behavior
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulties of inclusion of subjects
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1308093; 2013-A01352-43 (Other: ANSM)
Record Dates: First submitted 2015-09-11; First posted 2015-09-15 (Estimated); Last update posted 2021-11-17 (Actual); Status verified 2018-03

CONDITIONS: Pathological Gambler
Keywords: pathological gambler; Go-Nogo test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Gambler performing Go-Nogo (Experimental): In this study, Gambler performing Go-Nogo test. On a computer, various exercises (called "Go-Nogo") whose principle is: 2 symbols (for example, a circle and a square) appear in random order on the screen computer. The patient will not press the response button (key on the keyboard) that upon the occurrence of one of the two symbols, in dependence upon the command that it has been given by the psychiatrist, and this as quickly as possible. The patient will successively perform 3 versions of this exercise (with a neutral wallpaper, with neutral/games images or with neutral/games tones). Order of the 3 versions will be determined by randomization.
  Interventions: Other: Go-Nogo test
- Social layer performing Go-Nogo (Active Comparator): In this study, social player performing Go-Nogo test. On a computer, various exercises (called "Go-Nogo") whose principle is: 2 symbols (for example, a circle and a square) appear in random order on the screen computer. The patient will not press the response button (key on the keyboard) that upon the occurrence of one of the two symbols, in dependence upon the command that it has been given by the psychiatrist, and this as quickly as possible. The patient will successively perform 3 versions of this exercise (with a neutral wallpaper, with neutral/games images or with neutral/games tones). Order of the 3 versions will be determined by randomization.
  Interventions: Other: Go-Nogo test
- non-gamer witnesses performing Go-Nogo (Placebo Comparator): In this study, non-gamer witnesses performing Go-Nogo test. On a computer, various exercises (called "Go-Nogo") whose principle is: 2 symbols (for example, a circle and a square) appear in random order on the screen computer. The patient will not press the response button (key on the keyboard) that upon the occurrence of one of the two symbols, in dependence upon the command that it has been given by the psychiatrist, and this as quickly as possible. The patient will successively perform 3 versions of this exercise (with a neutral wallpaper, with neutral/games images or with neutral/games tones). Order of the 3 versions will be determined by randomization.
  Interventions: Other: Go-Nogo test

INTERVENTIONS:
Other: Go-Nogo test — In this study, Gambler performing Go-Nogo test. On a computer, various exercises (called "Go-Nogo") whose principle is: 2 symbols (for example, a circle and a square) appear in random order on the screen computer. The patient will not press the response button (key on the keyboard) that upon the occurrence of one of the two symbols, in dependence upon the command that it has been given by the psychiatrist, and this as quickly as possible. The patient will successively perform 3 versions of this exercise (with a neutral wallpaper, with neutral/games images or with neutral/games tones). Order of the 3 versions will be determined by randomization.

SUMMARY:
In France, the prevalence of problem gambling and risk has been estimated at 1.3%. This disorder, currently considered a behavioral addiction is characterized by a loss of control and an excessive focus on the game.

The literature on intervening psychological mechanisms in the development of the game led to think that the size of loss of control, central among players, could be understood as a reduction in control capacity but also as automatic activation behavior game.

The task of Go-Nogo, commonly used in cognitive psychology, assesses the automatic and controlled components of behavior. Furthermore, different models of the concept of addiction underline the importance of the environment associated with addiction. However, no study takes into account the interaction between the game environment and the involvement of these mechanisms.

DETAILED DESCRIPTION:
In this study, patients will realize, on a computer, various exercises (called "Go-Nogo") whose principle is: 2 symbols (for example, a circle and a square) appear in random order on the screen computer. The patient will not press the response button (key on the keyboard) that upon the occurrence of one of the two symbols, in dependence upon the command that it has been given by the psychiatrist, and this as quickly as possible. The patient will successively perform 3 versions of this exercise (with a neutral wallpaper, with neutral/games images or with neutral/games tones).Order of the 3 versions will be determined by randomization.

ELIGIBILITY:
Inclusion Criteria:

* For pathological gambler (JP): active casino players meet the diagnostic criteria for pathological gambling according to DSM-IV-TR
* For social player (JS): casino players who score the SOGS is less than or equal to 2, and playing at least once a month in a money game and chance.
* For non-gamer witnesses (T): play less than once per month to any type of gambling, except for Lotto and Euromillion where the threshold is increased at least once a week. These two draw games are considered more socially enrolled in a leisure practice without necessarily enroll in gambling.
* Right handed
* Aged between 18-60 years.
* Without psychotropic treatment or treatment with a stable and unchanged for over a month.

Exclusion Criteria:

* Participants with a problem of visual acuity and / or uncorrected hearing.
* Other current addiction (except tobacco, for reasons of feasibility).
* Current Psychiatric comorbidity
* Treatment psychotropic introduced or changed for less than a month.
* Subjects with atrial fibrillation, with a pacemaker and / or receiving antiarrhythmic drugs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2014-04-30 (Actual); Study Completion 2014-04-30 (Actual)

PRIMARY OUTCOMES:
Result Go-Nogo test | day 1
  Difference between the number of errors (control) in Go-Nogo test simple and visual-auditory Go-Nogo (composite measure)

CONTACTS AND LOCATIONS:
Overall Officials: Aurelia GAY, MD, Principal Investigator — CHU de SAINT-ETIENNE
Locations (1):
- CHU de SAINT-ETIENNE, Saint-Etienne, France